CLINICAL TRIAL: NCT04347304
Title: Effects of Flavanol-rich Dark Chocolate Consumption on Metabolic Profiles Among Obese
Brief Title: Effects of Flavanol-rich Dark Chocolate Consumption on Metabolic Profiles Among Obese Adults Using Metabolomics Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Hasmiza Halib, Principle Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-19-3092-51617.
Record Dates: First submitted 2020-04-07; First posted 2020-04-15 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: Obesity; Cocoa polyphenols; Dark chocolate
MeSH Terms: conditions — Obesity | interventions — Polyphenols

STUDY DESIGN:
Intervention Model Description: A randomized, open-labelled, parallel controlled trial will be conducted in Universiti Putra Malaysia from October 2021 until December 2022 involving obese adult aged 18 - 45 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cocoa polyphenols (Experimental): 21 grams of dark chocolate (289 mg polyphenols)
  Interventions: Dietary Supplement: Dark chocolate (20 grams) per day providing 508 mg of polyphenols
- polyphenols free (Placebo Comparator): 21 grams of white chocolate (0 mg polyphenols)
  Interventions: Dietary Supplement: white chocolate (20 grams) with no polyphenols

INTERVENTIONS:
Dietary Supplement: Dark chocolate (20 grams) per day providing 508 mg of polyphenols — subjects will be given 21 grams of dark chocolate providing 289 mg of polyphenols per day for 12 weeks.
  Arms: cocoa polyphenols
Dietary Supplement: white chocolate (20 grams) with no polyphenols — subjects will be given 21 grams of white chocolate (0 mg polyohenols) per day for 12 weeks
  Arms: polyphenols free

SUMMARY:
Obesity has become a global issue due to its alarming high and increasing prevalence worldwide and the roles it plays in occurrence of many chronic diseases. In addition, obesity is characterized as a state of chronic, low-grade inflammation and is associated with an abnormal inflammatory response, low antioxidant capacity and reduced insulin sensitivity which lead to the generation of inflammation, oxidative stress and insulin resistance.

As in Malaysia, study by National Health and Morbidity Survey Malaysia (NHMS) in 2011 and 2015 showed a continuing increase of the problem. In response to the rise of obesity prevalence, various efforts and strategies have been implemented in the past decade to combat this problem. The use of natural products as therapeutic agents in preventing metabolic disease has becoming popular. Cocoa and its products is a largely consumed food in the world. It has a very rich sources of phenolic compound. Several in vitro and in vivo studies have shown that polyphenols, with antioxidant, anti-inflammatory and anti-obesity properties, can boost energy expenditure and thermogenesis, lessen oxidative stress and inflammation while supporting weight loss management. Furthermore, the contribution of human studies especially among obese relatively limited.

The popularity of chocolate and/or cocoa and its frequent consumption made it the target of many research studies, due to its favourable effects, and to the significant role it may exert on improving the obesity condition. Therefore, this study aims to investigate the effects of flavanol-rich dark chocolate consumption on metabolic profiles of obese adults using metabolomic approach.

DETAILED DESCRIPTION:
Overnutrition and sedentary lifestyle are the leading factors associated with the development of obesity. Obese adults usually are advised to make lifestyle modifications which include dietary restriction and physical activity recommendation. In addition, dietary supplements and medication such as anti-hypertensive, lipid lowering drugs are used to achieved targeted body weight of obese adult. Therefore, the confounding factors in this study namely dietary intake, physical activity, medication, supplements were controlled throughout the study. These factors including smoking were also controlled as it will affect the metabolites.

Imbalance between energy intake and expenditure results in adipose tissue expansion due to excessive lipogenesis in adipose tissues. Generally, it is well accepted that adipose tissue expansion in an obese state is accompanied by elevated inflammation. Oxidative stress and pro-inflammatory processes are strongly related. Increased abdominal adipose tissue accelerates the production of pro-inflammatory cytokines which promote increased generation of ROS, both inflammation and oxidative stress play a significant role in the development of insulin resistant thus further are associated with the degree of metabolic dysfunction.

It was hypothesized that cocoa flavanol with the properties of anti-inflammation, anti-oxidative and antiobesity properties may reduce the oxidative stress and inflammation, subsequently reduce the insulin resistance and thus improved the outcome measurements in obese adult. In order to measures the altered metabolite in the urine and blood serum following cocoa rich flavanol consumption in dark chocolate in obese adult, a metabolomics based approach is used in this study.

This study is a randomized, open-labelled, parallel controlled trial where the intervention group will receive 20 grams of dark chocolate, daily for 12 weeks while the control group will receive 20 grams of white chocolate daily for 12 weeks. Measurement will be taken including sociodemographic, anthropometric measurement, diet and physical activity questionnaire, blood and urine samples at baseline and 12 weeks of intervention. Obese male adult aged 18-45 years old will be recruited

ELIGIBILITY:
Inclusion Criteria:

* Malaysian
* Obese BMI ≥ 25.0 kg/m2
* Not on any drug or herbal preparation, antioxidative or any drugs or dietary supplement.
* Do not have any chronic diseases
* Do not have allergy to cocoa
* Age 18-45 years old.

Exclusion Criteria:

* Non-Malaysian
* BMI < 25.0 kg/m2
* Smokers and alcohol drinkers
* Participants with cardiovascular diseases, hypertension or diabetes
* Participants taking medications that affect insulin, glucose, lipid or blood pressure levels
* Participants taking any dietary supplements
* Have allergy towards cocoa beverages
* Participants who are currently involved in a weight management program

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-03-23 (Estimated); Primary Completion 2022-06-23 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
change in insulin resistance at 12 week | baseline and 8 weeks
  Insulin resistance will be determined HOMA-IR and calculated as HOMA-IR = fasting serum x fasting blood glucose/22.5.
change in insulin sensitivity at 8 weeks | baseline and 8 weeks
  To assess insulin sensitivity, Quantitative Insulin Sensitivity Check Index (QUICKI) will be used and cutt off point of less than 0.33 indicates reduced insulin sensitivity

SECONDARY OUTCOMES:
change in body weight at 8 weeks | baseline and 8 weeks
  Body weight will be measured in kilograms using SECA electronic scale model 703.
change in waist circumference at 8 weeks | baseline and 8 weeks
  Waist circumference will be assessed at the midpoint between the lowest rib andd the iliac crest using a non-stretchable tape measure. The measurement will be conducted twice to the nearest 0.1cm. The cutoff points for waist ciircumference by WHO expert committee on obesity in Asian and Pacific populations are >90 cm for men and >80cm fro women.
change in lipid profiles (TG, HDL-c, LDL-c, TC) at 8 weeks | baseline and 8 weeks
  Lipid profiles (TG, Cholesterol, LDL-c, and HDL-c) will be determined using commercially available kits using Architect ci8200 analyzer
change in inflammatory markers (C-reactive protein ) at 8 week | baseline and 8 weeks
  C-reactive protein will be measured using kits of human inflammatory cytokines by Enzyme Linked Inmuno Sorbent Assay from blood serum and will be expressed as mg/L.
change in oxidative stress markers (oxidized LDL) at 8 week | baseline and 8 weeks
  Levels of LDL-ox in plasma will be analysed at the beginning and the end (8 weeks) and will be expressed as mg/L.
changes in metabolomics profiles following flavanol-rich dark chocolate consumption at 8 week | baseline and 8 weeks
  Metabolomic analysis of the plasma sample will be performed using 1H-NMR platform
changes in gut microbiome status following flavanol-rich dark chocolate consumption at 8 week | baseline and 8 weeks
  metagenomic analysis of fecal samples will be analysed at the beginning and end (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Amin Ismail, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Seri Kembangan, Selangor, Malaysia

REFERENCES:
- [Background] Moazzami AA, Bondia-Pons I, Hanhineva K, Juntunen K, Antl N, Poutanen K, Mykkanen H. Metabolomics reveals the metabolic shifts following an intervention with rye bread in postmenopausal women--a randomized control trial. Nutr J. 2012 Oct 22;11:88. doi: 10.1186/1475-2891-11-88. PMID 23088297
- [Background] Hensley K, Robinson KA, Gabbita SP, Salsman S, Floyd RA. Reactive oxygen species, cell signaling, and cell injury. Free Radic Biol Med. 2000 May 15;28(10):1456-62. doi: 10.1016/s0891-5849(00)00252-5. PMID 10927169
- [Background] Suhre K, Meisinger C, Doring A, Altmaier E, Belcredi P, Gieger C, Chang D, Milburn MV, Gall WE, Weinberger KM, Mewes HW, Hrabe de Angelis M, Wichmann HE, Kronenberg F, Adamski J, Illig T. Metabolic footprint of diabetes: a multiplatform metabolomics study in an epidemiological setting. PLoS One. 2010 Nov 11;5(11):e13953. doi: 10.1371/journal.pone.0013953. PMID 21085649